CLINICAL TRIAL: NCT01964430
Title: A Phase 3, Multicenter, Open-label, Randomized Study of Nab-Paclitaxel Plus Gemcitabine Versus Gemcitabine Alone as Adjuvant Therapy in Subjects With Surgically Resected Pancreatic Adenocarcinoma
Brief Title: Nab-paclitaxel and Gemcitabine vs Gemcitabine Alone as Adjuvant Therapy for Patients With Resected Pancreatic Cancer (the "Apact" Study)
Acronym: apact
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-PANC-003; 2013-003398-91 (EudraCT Number)
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Endocrine Gland Neoplasms; Pancreatic Diseases; Digestive System Diseases; Endocrine System Diseases; Gemcitabine; Antimetabolites, Antineoplastic
Keywords: Resectable pancreatic cancer; resected; resectable PDA; adenocarcinoma; surgically resected; adjuvant; Abraxane; nab-paclitaxel; ABI-007; gemcitabine; Gemzar; Phase 3
MeSH Terms: conditions — Pancreatic Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Endocrine Gland Neoplasms; Pancreatic Diseases; Digestive System Diseases; Endocrine System Diseases; Adenocarcinoma | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nab-Paclitaxel 125 mg/m^2 plus gemcitabine 1000 mg/m2 (Experimental): Participants received nab-Paclitaxel 125 mg/m^2 administered as an intravenous (IV) infusion over 30 to 40 minutes, followed by gemcitabine 1000 mg/m^2 as an IV infusion over 30 to 40 minutes on Days 1, 8 and 15 of each 28-day treatment cycle for 6 cycles, unless there was evidence of radiologic disease recurrence, unacceptable toxicity, subject or physician decision, withdrawal of consent, or death.
  Interventions: Drug: nab-Paclitaxel; Drug: Gemcitabine
- Gemcitabine 1000 mg/m^2 (Active Comparator): Participants received gemcitabine 1000 mg/m^2 administered as an IV infusion over 30 to 40 minutes on Days 1, 8 and 15 of each 28-day treatment cycle for 6 cycles, unless there was evidence of radiologic disease recurrence, unacceptable toxicity, subject or physician decision, withdrawal of consent, or death.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: nab-Paclitaxel — nab-Paclitaxel 125 mg/m^2 on Days 1, 8, and 15 of every 28 day treatment cycle by intravenous (IV) administration for a total of 6 cycles.
  Other Names: Abraxane
  Arms: nab-Paclitaxel 125 mg/m^2 plus gemcitabine 1000 mg/m2
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 on Days 1, 8, and 15 of a 28 day cycle by IV administration for a total of 6 cycles.
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to compare whether there is a delay or prevention of recurrence or death in participants with surgically removed pancreatic cancer who then take nab-Paclitaxel in combination with gemcitabine compared to those who take gemcitabine alone.

DETAILED DESCRIPTION:
ABI-007-PANC-003 is a Phase 3, international, multicenter, randomized, open-label, controlled study that will compare the efficacy of nab-paclitaxel in combination with gemcitabine to gemcitabine alone as adjuvant treatment for 6 cycles in patients with surgically resected pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed resected ductal pancreatic adenocarcinoma with macroscopic complete resection (R0 and R1). Subjects with neuroendocrine (and mixed type) tumors are excluded.
2. Pancreatic cancer surgical staging: Tumor (T) 1-3, Lymph Node (LN) N0-1, Metastasis (M) 0.
3. Subject should be able to start treatment no later than 12 weeks postsurgery.
4. ≥18 years of age at the time of signing the informed consent form (ICF).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Acceptable hematology parameters:

   * Absolute neutrophil count (ANC) ≥1500 cell/mm^3
   * Platelet count ≥100,000/mm^3
   * Hemoglobin (Hgb) ≥9 g/dL
7. Acceptable blood chemistry levels:

   * Aspartate aminotransferase (AST)/ serum glutamic oxaloacetic transaminase (SGOT) and alanine transaminase (ALT)/ serum glutamic -pyruvic transaminase (SGPT) ≤2.5 × upper limit of normal range (ULN)
   * Total bilirubin ≤ upper limit of normal (participants with Gilbert's syndrome can have bilirubin of up to 1.5 x ULN)
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Serum creatinine within upper limits of normal or calculated clearance ≥50 mL/min/1.73 m^2. If using creatinine clearance, actual body weight should be used for calculating creatinine clearance (eg, using the Cockroft-Gault formula). For subjects with a body mass index (BMI) >30 kg/m2, lean body weight should be used instead
8. Cancer antigen (CA)19-9 <100 U/mL assessed within 14 days of randomization
9. Acceptable coagulation studies as demonstrated by prothrombin time (PT) and partial thromboplastin time (PTT) within normal limits (±15%)

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Prior neo-adjuvant treatment or radiation therapy for pancreatic adenocarcinoma
2. Presence of or history of metastatic pancreatic adenocarcinoma
3. Any other malignancy within 5 years prior to randomization, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, or nonmelanomatous skin cancer (all treatment of which should have been completed 6 months prior to randomization)
4. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment
5. Known infection with hepatitis B or C, or history of human immunodeficiency virus (HIV) infection, or subject receiving immunosuppressive or myelosuppressive medications that would in the opinion of the investigator, increase the risk of serious neutropenic complications
6. History of allergy or hypersensitivity to nab-paclitaxel or gemcitabine or any of their excipients
7. Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the subject's safety or the study data integrity. These include, but are not limited to:

   1. History of connective tissue disorders (eg, lupus, scleroderma, arteritis nodosa)
   2. History of interstitial lung disease, slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies
   3. History of the following within 6 months prior to Cycle 1 Day 1: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or electrocardiogram (ECG) abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 866 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (341):
- United States (107):
  - Local Institution - 043, Scottsdale, Arizona
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - UCSD Moores Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Local Institution - 044, Sacramento, California
  - UC Davis Cancer Center, Sacramento, California
  - Local Institution - 001, San Francisco, California
  - University of California, San Francisco Cutaneous Oncology and Melanoma Center, San Francisco, California
  - University of California Los Angeles, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Local Institution - 059, Denver, Colorado
  - Rocky Mountain Cancer Centers, LLP [Denver-Midtown], Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Local Institution - 022, Boca Raton, Florida
  - Lynn Cancer Institute, Boca Raton, Florida
  - Florida Cancer Institute Cancer Spec, Fort Myers, Florida
  - Local Institution - 031, Fort Myers, Florida
  - Gainesville Heme Oncology Associates, Gainesville, Florida
  - Local Institution - 011, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - University of Miami and Sylvester Cancer Center, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Local Institution - 039, Orlando, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Georgia Cancer Specialist, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Northshore University Healthsystem Research Institute, Evanston, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Ochsner Medical Center - Jefferson Highway, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel-Deaconess Medical Center, Boston, Massachusetts
  - Local Institution - 040, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - 045, Boston, Massachusetts
  - Local Institution - 036, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Center Wayne State University, Detroit, Michigan
  - Local Institution - 021, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Local Institution - 048, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Local Institution - 064, Basking Ridge, New Jersey
  - MSKCC Basking Ridge, Basking Ridge, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Local Institution - 025, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center West Harrison, Harrison, New York
  - NYU Langone Medical Center, Lake Success, New York
  - Local Institution - 008, New York, New York
  - Memorial Sloan-Kettering Cancer Center - NYC, New York, New York
  - Columbia University Medical Center, New York, New York
  - Local Institution - 032, New York, New York
  - Local Institution - 013, Rochester, New York
  - University of Rochester Cancer Center, James P. Wilmot Cancer Center, Rochester, New York
  - Local Institution - 066, Rockville Centre, New York
  - MSKCC at Mercy Medical Center Mercy RockvilleCenter, Rockville Centre, New York
  - MSKCC at Phelps Memorial Hospital Center. Phelps Sleepy Hollow, Sleepy Hollow, New York
  - State University of New York Upstate Medical Center, Syracuse, New York
  - Local Institution - 051, Winston-Salem, North Carolina
  - Wake Forest Univ. Health Sciences Outpatient Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Local Institution - 030, Cincinnati, Ohio
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - University of Cincinnati Medical CenterDivsion of Hematology OncologyThe Barrett Center, Cincinnati, Ohio
  - Case Western Reserve Center, Cleveland, Ohio
  - Local Institution - 047, Cleveland, Ohio
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Cleveland Clinic Foundation IRB, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Local Institution - 020, Cleveland, Ohio
  - Local Institution - 054, Cleveland, Ohio
  - Local Institution - 005, Columbus, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Local Institution - 049, Oklahoma City, Oklahoma
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Local Institution - 019, Portland, Oregon
  - Oregon Health and Science University OHSU, Portland, Oregon
  - Local Institution - 016, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Local Institution - 027, Pittsburgh, Pennsylvania
  - UPMC Cancer Pavillion, Pittsburgh, Pennsylvania
  - Chattanooga Oncology Hematology Care, Chattanooga, Tennessee
  - Local Institution - 023, Chattanooga, Tennessee
  - Local Institution - 004, Nashville, Tennessee
  - Sarah Cannon Research Inst, Nashville, Tennessee
  - Local Institution - 002, Nashville, Tennessee
  - Vanderbilt- Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Baylor Sammons Cancer Center, Dallas, Texas
  - Local Institution - 062, Dallas, Texas
  - Local Institution - 010, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Local Institution - 050, Fort Worth, Texas
  - The Center for Cancer and Blood Disorders - Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Local Institution - 041, Houston, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Local Institution - 038, Charlottesville, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Local Institution - 003, Seattle, Washington
  - Seattle Cancer Care Alliance - Seattle, Seattle, Washington
  - Virginia Mason Cancer Center, Seattle, Washington
  - Local Institution - 014, Madison, Wisconsin
  - University of Wisconsin - Madison Cancer Center, Madison, Wisconsin
- Australia (21):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Local Institution - 505, Garran, Australian Capital Territory
  - Local Institution - 501, Darlinghurst, New South Wales
  - Local Institution - 507, St Leonards, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Local Institution - 504, Herston, Queensland
  - ICON Cancer Center, Milton, Queensland
  - Local Institution - 502, Milton, Queensland
  - Local Institution - 506, Bentleigh East, Victoria
  - Local Institution - 508, Subiaco, Western Australia
  - St John of God Subiaco Hospital, Subiaco, Western Australia
  - Monash Medical Centre Moorabbin Campus, Bentleigh East
  - Saint Vincent's Hospital, Darlinghurst
  - Austin Hospital, Heidelberg
  - Local Institution - 509, Heidelberg
  - Royal Brisbane and Women's Hospital, Herston
  - Cabrini Hospital, Malvern
  - Local Institution - 503, Malvern
  - Local Institution - 500, Randwick
  - Prince of Wales Hospital, Randwick
  - The Queen Elizabeth Hospital, Woodville South
- Austria (16):
  - Local Institution - 205, Graz
  - Medical University of Graz, Graz
  - Local Institution - 203, Innsbruck
  - Medical University Innsbruck, Innsbruck
  - Hospital of Elisabethinen Linz, Linz
  - Local Institution - 206, Linz
  - Local Institution - 204, Salzburg
  - Salzburger Landkliniken St. Johanns-Spital, Salzburg
  - Local Institution - 200, Vienna
  - Medizinische Universitat Wien, Vienna
  - Kaiser-Franz-Josef Spital, Vienna
  - Local Institution - 201, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
  - Local Institution - 0207, Wels
  - Hospital Wiener Neustadt, Wiener Neustadt
  - Local Institution - 202, Wiener Neustadt
- Belgium (7):
  - Hopital Erasme, Brussels
  - Local Institution - 211, Brussels
  - UZ Antwerpen, Edegem
  - Local Institution - 213, Ghent
  - UZ Gent, Ghent
  - Local Institution - 210, Leuven
  - UZ Leuven, Leuven
- Canada (10):
  - Local Institution - 102, Calgary, Alberta
  - Tom Baker Cancer Center, Calgary, Alberta
  - Local Institution - 101, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Local Institution - 100, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de L'Universite de Montreal St-Luc, Montreal, Quebec
  - Local Institution - 104, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Local Institution - 103, Montreal, Quebec
- Czechia (5):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Local Institution - 220, Hradec Králové
  - Krajska nemocnice Liberec, a.s., Liberec
  - Krajska nemocnice T. Bati a.s., Zlín
  - Local Institution - 221, Zlín
- Denmark (6):
  - Hæmatologisk afd. B Aalborg Sygehus Syd, Aalborg
  - Local Institution - 231, Aalborg
  - Herlev Hospital, Herlev
  - Local Institution - 232, Herlev
  - Local Institution - 230, Odense C
  - Onk.Dep., Odense Universitets hospital, Odense C
- Finland (6):
  - Local Institution - 240, Tampere, Oulun Lääni
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Local Institution - 241, Helsinki
  - Tampereen yliopistollinen sairaala, Tampere
  - Local Institution - 242, Turku
  - Turku University Hospital, Turku
- France (18):
  - Center Hospitalier Universitaire d' Angers, Angers
  - Local Institution - 253, Angers
  - Hopital Henri Mondor, Créteil
  - CHRU de Lille France, Lille
  - Local Institution - 257, Lille
  - Hopital prive Jean Mermoz, Lyon
  - Local Institution - 252, Lyon
  - Hopital Edouard Herriot - Hepato-gastroenterologie, Lyon
  - Local Institution - 258, Lyon
  - Hopital Europeen Georges Pompidou, Paris
  - Local Institution - 250, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Pitie Salpetriere, Paris
  - Local Institution - 259, Paris
  - CHU La Miletrie, Poitiers
  - Local Institution - 251, Poitiers
  - Local Institution - 256, Toulose
  - Pole Des Specialites Medicales, Hopital Purpan, Toulose
- Germany (31):
  - Klinikum Weiden, Bayern
  - Local Institution - 280, Bayern
  - Charite - Universitätsmedizin Berlin, Berlin
  - Local Institution - 272, Berlin
  - Local Institution - 281, Cologne
  - Praxis Internistischer Onkologie und Hamatologie Koln, Cologne
  - Local Institution - 278, Dresden
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Kliniken Essen-Mitte, Essen
  - Local Institution - 277, Frankfurt
  - Universitatsklinkum Frankfurt, Frankfurt
  - Local Institution - 284, Frechen
  - Praxis Internistischer Onkologie und Hamatologie Frechen, Frechen
  - Local Institution - 275, Friedrichshafen
  - Praxis für Innere Medizin, Dr.Oettle Helmut, Friedrichshafen
  - Ernst-Moritz-Arndt-Universität Greifswald, Greifswald
  - Local Institution - 279, Greifswald
  - Local Institution - 273, Hamburg
  - Universitaetsklinik Hamburg - Eppendorf, Hamburg
  - Local Institution - 274, Magdeburg
  - Universitatsklinik Magdeburg, Magdeburg
  - Klinikum der Johannes Gutenberg Uniervsitaet ,Haematologie, Mainz
  - Local Institution - 283, Mainz
  - Klinikum der Universitat Munchen-Grosshadern, München
  - Local Institution - 282, München
  - Klinikum Neuperlach, München
  - Local Institution - 276, München
  - Local Institution - 0271, Tübingen
  - University of Tubingen, Tübingen
  - Local Institution - 270, Würzburg
  - Universitatsklinikum Würzburg, Würzburg
- Hong Kong (5):
  - Local Institution - 601, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Local Institution - 602, Shatin
  - Prince of Wales Hospital the Chinese University of Hong Kong, Shatin
- Hungary (11):
  - Fovarosi Szent Istvan es Szent Laszlo Korhaz es Rendelointezet, Budapest
  - Local Institution - 293, Budapest
  - Local Institution - 291, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Local Institution - 290, Debrecen
  - Local Institution - 292, Győr
  - Petz Aladar Megyei Oktato Korhaz,II. Belgyogyaszat, Győr
  - Local Institution - 295, Szeged
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Szent-Gyorgyi Albert TE AOK Borgyogy, Szeged
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Ireland (4):
  - Local Institution - 311, Cork
  - Cork University Hospital, Cork
  - Local Institution - 310, Dublin
  - St Vincent's University Hospital, Dublin
- Italy (28):
  - Local Institution - 329, Terni, Umbria
  - Local Institution - 325, Ancona
  - Ospedali Riuniti Umberto I GM Lancisi, Ancona
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Local Institution - 330, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Local Institution - 328, Florence
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori (I.R.S.T.), Meldola
  - Local Institution - 331, Meldola
  - Local Institution - 321, Milan
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliera Niguarda Ca Granda, Milan
  - Local Institution - 322, Milan
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Local Institution - 324, Pisa
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Local Institution - 333, Reggio Emilia
  - Local Institution - 323, Roma
  - Local Institution - 327, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Local Institution - 326, Rozzano (MI)
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Local Institution - 332, San Giovanni Rotondo
  - Azienda Ospedaliera S Maria di Terni, Terni
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
  - Local Institution - 320, Verona
- Netherlands (6):
  - Academisch Medisch Centrum Amsterdam, Amsterdam
  - Local Institution - 400, Amsterdam
  - Catharina Hospital, Eindhoven
  - Local Institution - 403, Eindhoven
  - Isala Klinieken, Zwolle
  - Local Institution - 402, Zwolle
- Portugal (6):
  - Centro Hospitalar de Lisboa Central - Hospital de Santo António dos Capuchos, Lisbon
  - Local Institution - 340, Lisbon
  - Hospital Da Luz, Lisbon
  - Local Institution - 341, Lisbon
  - Hospital de Sao Joao, Porto
  - Local Institution - 342, Porto
- Singapore (4):
  - Local Institution - 610, Singapore
  - National University Hospital, Singapore
  - Local Institution - 611, Singapore
  - National Cancer Center, Singapore
- South Korea (6):
  - Local Institution - 641, Seoul
  - Seoul National University Hospital, Seoul
  - Local Institution - 642, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Local Institution - 640, Seoul
- Spain (26):
  - Local Institution - 371, Santander, Cantabria
  - Local Institution - 360, Barcelona
  - Clinic Barcelona Hospital Universitari, Barcelona
  - Local Institution - 363, Barcelona
  - Instituto Catalan de Oncologia-Hospital Duran, Barcelona
  - Local Institution - 370, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Gregorio Maranon, Madrid
  - Local Institution - 367, Madrid
  - Local Institution - 362, Madrid
  - Ramon y Cajal Univeresity Hospital, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Local Institution - 372, Madrid
  - Hospital 12 de Octubre, Madrid
  - Local Institution - 365, Madrid
  - Centro Integral, Madrid
  - Local Institution - 361, Madrid
  - Hospital General Carlos Haya, Málaga
  - Local Institution - 369, Málaga
  - Complejo Hospitalario de Navarra, Pamplona/ Navarra
  - Local Institution - 368, Pamplona/ Navarra
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario De Santiago De Compostela, Santiago de Compostela
  - Local Institution - 366, Santiago de Compostela
  - Hospital Virgen del Rocio, Seville
  - Local Institution - 364, Seville
- Taiwan (12):
  - Local Institution - 620, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Local Institution - 625, Tainan, Taiana
  - National Cheng Kung University Hospital, Tainan, Taiana
  - Local Institution - 623, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Local Institution - 622, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
  - Local Institution - 624, Taoyuan District
  - Local Institution - 621, Tapei
  - National Taiwan University Hospital, Tapei
- United Kingdom (6):
  - Addenbrookes Hospital, Cambridge
  - Local Institution - 382, Cambridge
  - Glasgow Royal Infirmary, Glasgow
  - Local Institution - 380, Glasgow
  - Local Institution - 381, Sheffield
  - Weston Park Hospital, Sheffield South Yorkshire

REFERENCES:
- [Background] Young R, Mainwaring P, Clingan P, Parnis FX, Asghari G, Beale P, Aly A, Botteman M, Romano A, Ferrara S, Margunato-Debay S, Harris M. nab-Paclitaxel plus gemcitabine in metastatic pancreatic adenocarcinoma: Australian subset analyses of the phase III MPACT trial. Asia Pac J Clin Oncol. 2018 Oct;14(5):e325-e331. doi: 10.1111/ajco.12999. Epub 2018 Jun 22. PMID 29932294
- [Background] Reni M, Zanon S, Balzano G, Passoni P, Pircher C, Chiaravalli M, Fugazza C, Ceraulo D, Nicoletti R, Arcidiacono PG, Macchini M, Peretti U, Castoldi R, Doglioni C, Falconi M, Partelli S, Gianni L. A randomised phase 2 trial of nab-paclitaxel plus gemcitabine with or without capecitabine and cisplatin in locally advanced or borderline resectable pancreatic adenocarcinoma. Eur J Cancer. 2018 Oct;102:95-102. doi: 10.1016/j.ejca.2018.07.007. Epub 2018 Aug 24. PMID 30149366
- [Background] Fernandez A, Salgado M, Garcia A, Buxo E, Vera R, Adeva J, Jimenez-Fonseca P, Quintero G, Llorca C, Canabate M, Lopez LJ, Munoz A, Ramirez P, Gonzalez P, Lopez C, Reboredo M, Gallardo E, Sanchez-Canovas M, Gallego J, Guillen C, Ruiz-Miravet N, Navarro-Perez V, De la Camara J, Ales-Diaz I, Pazo-Cid RA, Carmona-Bayonas A. Prognostic factors for survival with nab-paclitaxel plus gemcitabine in metastatic pancreatic cancer in real-life practice: the ANICE-PaC study. BMC Cancer. 2018 Nov 29;18(1):1185. doi: 10.1186/s12885-018-5101-3. PMID 30497432
- [Background] Sonbol MB, Ahn DH, Goldstein D, Okusaka T, Tabernero J, Macarulla T, Reni M, Li CP, O'Neil B, Van Cutsem E, Bekaii-Saab T. CanStem111P trial: a Phase III study of napabucasin plus nab-paclitaxel with gemcitabine. Future Oncol. 2019 Apr;15(12):1295-1302. doi: 10.2217/fon-2018-0903. Epub 2019 Feb 15. PMID 30768369
- [Derived] Tempero MA, Pelzer U, O'Reilly EM, Winter J, Oh DY, Li CP, Tortora G, Chang HM, Lopez CD, Bekaii-Saab T, Ko AH, Santoro A, Park JO, Noel MS, Frassineti GL, Shan YS, Dean A, Riess H, Van Cutsem E, Berlin J, Philip P, Moore M, Goldstein D, Tabernero J, Li M, Ferrara S, Le Bruchec Y, Zhang G, Lu B, Biankin AV, Reni M; APACT Investigators. Adjuvant nab-Paclitaxel + Gemcitabine in Resected Pancreatic Ductal Adenocarcinoma: Results From a Randomized, Open-Label, Phase III Trial. J Clin Oncol. 2023 Apr 10;41(11):2007-2019. doi: 10.1200/JCO.22.01134. Epub 2022 Dec 15. PMID 36521097
- [Derived] Reni M, Braverman J, Hendifar A, Li CP, Macarulla T, Oh DY, Riess H, Tempero M, Lu B, Marcus J, Joshi N, Botteman M, Dueck AC. Evaluation of Minimal Important Difference and Responder Definition in the EORTC QLQ-PAN26 Module for Assessing Health-Related Quality of Life in Patients with Surgically Resected Pancreatic Adenocarcinoma. Ann Surg Oncol. 2021 Nov;28(12):7545-7554. doi: 10.1245/s10434-021-09816-z. Epub 2021 Apr 3. PMID 33813673
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study randomized participants at 160 sites in 21 countries: Australia, Austria, Belgium, Canada, Czech Republic, Denmark, Finland, France, Germany, Hong Kong, Hungary, Ireland, Italy, Netherlands, Portugal, Singapore, Republic of Korea, Spain, Taiwan, United Kingdom and the US.
Pre-assignment Details: Participants were randomized using a stratified randomization with a 1:1 ratio to either nab-paclitaxel followed by gemcitabine, or gemcitabine alone. Stratification factors were tumor resection status (R0 versus R1), nodal status lymph node positive versus lymph node negative, and region [North America, Europe, and Australia versus Asia Pacific]).
Groups:
- Nab-Paclitaxel and Gemcitabine: Participants received nab-Paclitaxel 125 mg/m^2 administered as an intravenous (IV) infusion over 30 to 40 minutes, followed by gemcitabine 1000 mg/m^2 as an IV infusion over 30 to 40 minutes on Days 1, 8 and 15 of each 28-day treatment cycle for 6 cycles, unless there was evidence of radiologic disease recurrence, unacceptable toxicity, participant or physician decision, withdrawal of consent, or death.
- Gemcitabine: Participants received gemcitabine 1000 mg/m^2 administered as an IV infusion over 30 to 40 minutes on Days 1, 8 and 15 of each 28-day treatment cycle for 6 cycles, unless there was evidence of radiologic disease recurrence, unacceptable toxicity, participant or physician decision, withdrawal of consent, or death.
Period: Pre-Treatment (Randomization) Period
Arm/Group | Nab-Paclitaxel and Gemcitabine | Gemcitabine
Started | 432 | 434
Completed (Participants continuing to Treatment) | 429 | 423
Not Completed | 3 | 11
Not completed — Protocol Deviation | 0 | 2
Not completed — Withdrawal by Subject | 2 | 9
Not completed — Adverse Event | 1 | 0
Period: Treatment Period
Arm/Group | Nab-Paclitaxel and Gemcitabine | Gemcitabine
Started | 429 | 423
Completed | 287 | 310
Not Completed | 142 | 113
Not completed — Adverse Event | 71 | 37
Not completed — Withdrawal by Subject | 36 | 27
Not completed — Death | 1 | 3
Not completed — Protocol Deviation | 0 | 1
Not completed — Physician Decision | 5 | 4
Not completed — Disease Relapse | 28 | 38
Not completed — Other reasons | 1 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population consisted of all randomized participants regardless of whether the participant received any investigational product (IP) or had any efficacy assessments collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nab-Paclitaxel and Gemcitabine | Gemcitabine | Total
Number analyzed (Participants) | 432 | 434 | 866
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (9.58) | 62.9 (8.84) | 63.2 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 181 | 385
  Male | 228 | 253 | 481
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 15 | 26
  Not Hispanic or Latino | 400 | 393 | 793
  Unknown or Not Reported | 21 | 26 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 60 | 56 | 116
  Black or African American | 4 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  White | 333 | 339 | 672
  Other | 11 | 6 | 17
  Not Collected or Reported | 24 | 22 | 46
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 144 | 156 | 300
  Europe | 203 | 205 | 408
  Australia | 30 | 20 | 50
  Asia Pacific | 55 | 53 | 108
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m²] | 1.77 (0.226) | 1.78 (0.221) | 1.78 (0.224)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 to 5: 0 = Fully active, no restrictions; 1 = Restricted activity but ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities; 3 = Limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled, no self-care, confined to bed or chair; 5 = Dead
  Participants
    0 = Fully Active | 252 | 268 | 520
    1 = Restricted but Ambulatory | 180 | 166 | 346
    2 = Ambulatory but Unable to Work | 0 | 0 | 0
    3 = Limited Self-care | 0 | 0 | 0
    4 = Completely Disabled | 0 | 0 | 0
Physician Assessment of Peripheral Neuropathy [Count of Participants; unit: Participants] — Physician assessment for grading of peripheral neuropathy in participants receiving chemotherapy according to National Cancer Institute Common Toxicity Criteria (NCICTC): - Grade 1 = Asymptomatic: loss of deep tendon reflexes or paresthesia; - Grade 2 = Moderate symptoms: limiting instrumental Activities of Daily Living (ADLs); - Grade 3 = Severe symptoms: limiting self-care ADL; assistance device indicated; - Grade 4 = Life-threatening consequences: urgent intervention indicated.
  Participants
    Grade 0 | 404 | 408 | 812
    Grade 1 | 26 | 21 | 47
    Grade 2 | 0 | 1 | 1
    Grade 3 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0
    Missing | 2 | 4 | 6
Time from Surgery to Randomization [Median (Full Range); unit: Days] | 57.0 [23.0 to 90.0] | 56.0 [17.0 to 88.0] | 57.0 [17.0 to 90.0]
TNM Classification [Count of Participants; unit: Participants] — The TNM system is the most widely used cancer staging system. Most hospitals and medical centers use the TNM system as their main method for cancer reporting. In the TNM system: The T refers to the size and extent of the main tumor. The main tumor is usually called the primary tumor and the "T" followed by a number shows the size of the tumor. The N refers to the number of nearby lymph nodes that have cancer. The M refers to whether the cancer has metastasized. This means that the cancer has spread from the primary tumor to other parts of the body.
  Participants
    T1 = Tumor is 2 cm or smaller | 16 | 13 | 29
    T2 = Tumor is > 2 cm, but not larger than 5 cm | 38 | 37 | 75
    T3 = Tumor is larger than 5 cm | 377 | 384 | 761
    T4 = Tumor is any size, but has spread | 1 | 0 | 1
Nodal Status [Count of Participants; unit: Participants] — The nodal status refers to the N and includes the number of nearby lymph nodes that are positive or negative for cancer.
  Participants
    Lymph Node Positive (LN+) | 311 | 312 | 623
    Lymph Node Negative (LN-) | 121 | 122 | 243
Resection Status [Count of Participants; unit: Participants] — Resection status was based on investigational site data (pathology reports were collected, but central pathology review and/or standardization was not conducted).
  Participants
    R0 (tumor-negative resection margin) | 327 | 334 | 661
    R1 (tumor- positive resection margin) | 105 | 100 | 205

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimate for Disease Free Survival (DFS) According to the Independent Radiological Review Committee
Description: Disease free survival was defined as the time from the date of randomization to the date of disease recurrence or death, whichever occurred earlier. Disease recurrence was determined by the independent radiological review of computed tomography (CT) or magnetic resonance imaging (MRI) scans. Participants who did not have disease recurrence or did not die were censored at the last tumor assessment date with disease-free status or the randomization date if the last tumor assessment with disease-free status was missing. Disease-free status referred to a status that was neither being disease recurrent nor indeterminate or not evaluable. Participants who received new anti-cancer therapy or cancer-related surgery prior to disease recurrence or death were censored at the date of last tumor assessment with disease-free status prior to the start of new anti-cancer therapy or cancer-related surgery or the randomization date.
Time Frame: Date of randomization up to data cut off date of 31 December 2018; median DFS follow-up time for censored participants was 22.242 months for nab-Paclitaxel and gemcitabine and 13.832 months for gemcitabine alone
Population: The intent-to-treat population consisted of all randomized participants regardless of whether they received any investigational product (IP) or had any efficacy assessment collected.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel and Gemcitabine | Gemcitabine
Number analyzed (Participants) | 432 | 434
months | 19.4 [16.62 to 21.91] | 18.8 [13.83 to 20.30]
Statistical Analysis 1: Comparison: Nab-Paclitaxel and Gemcitabine vs Gemcitabine; Test type: Superiority; p = 0.1824, Log Rank; Stratified by resection status (R0 versus R1) and nodal status (LN+ versus LN); Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.729 to 1.063] — Estimated using stratified Cox proportional hazards model adjusting for strata of resection status (R0 versus R1) and nodal status (LN+ versus LN-)

2. Secondary Outcome: Kaplan Meier Estimate of Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization to the date of death. Participants who were alive at the end of study or clinical data cut were censored on the last-known-to-be-alive date or the clinical cutoff date, whichever was earlier.
Time Frame: From randomization to date of death; median OS follow-up time for censored participants was 77.832 months for nab-Paclitaxel and gemcitabine and 77.799 months for gemcitabine alone
Population: The intent-to-treat population consisted of all randomized participants regardless of whether the participant received any IP or had any efficacy assessment collected.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel and Gemcitabine | Gemcitabine
Number analyzed (Participants) | 432 | 434
months
  25th Quartile | 20.7 [19.38 to 22.83] | 17.7 [14.78 to 19.91]
  50th Quartile | 41.8 [35.55 to 47.28] | 37.7 [31.11 to 40.51]
  75th Quartile | 90.2 [83.55 to NA] — Insufficient number of participants with events | 83.0 [61.93 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Nab-Paclitaxel and Gemcitabine vs Gemcitabine; Test type: Superiority; p = 0.0128, Log Rank; Stratified by resection status (R0 versus. R1) and nodal status (LN+ versus. LN-); Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.691 to 0.957] — Estimated using stratified Cox proportional hazards model adjusting for strata of resection status (R0 versus R1) and nodal status (LN+ versus

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE's)
Description: TEAEs are defined as any adverse event (AE) that begin or worsen on or after the start of study drug or procedure of the study period through the maximum duration of the period plus 28 days. The severity of AEs was graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 and the scale: Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death. Relation to study drug was determined by the investigator. A treatment-related TEAE is defined as TEAE which was considered to be related to one or both of the study drugs and reported as 'Suspected' on the case report form. AEs with a missing relationship were treated as 'treatment-related' in data summaries. IP (investigational product) refers to nab-Paclitaxel and/or Gemcitabine. "Related" TEAE refers to relation to study drug (IP).
Time Frame: From day 1 of study drug up to 28 days after the last dose of study drug; up to the data cut off date of 31 December 2018 (up to approximately 37 weeks).
Population: Treated Population consisted of randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel and Gemcitabine | Gemcitabine
Number analyzed (Participants) | 429 | 423
Participants
  ≥1 TEAE | 429 | 417
  ≥1 Related TEAE | 423 | 399
  ≥1 TEAE of Severity Grade 3 or Higher | 371 | 286
  ≥ 1 Related TEAE of Severity Grade 3 or Higher | 332 | 239
  ≥1 Serious TEAE | 176 | 96
  ≥1 Serious Related TEAE | 102 | 55
  ≥1 TEAE Leading to Withdrawal of IP | 117 | 43
  ≥1 Related TEAE Leading to Withdrawal of IP | 98 | 35
  ≥1 TEAE Lead Dose Reduction: nab-Paclitaxel or Gem | 276 | 210
  ≥1 Related TEAE Dose Reduct: nab-Paclitaxel or Gem | 270 | 205
  TEAE Lead Dose Interruption nab-Paclitaxel or Gem | 266 | 158
  ≥1 Related TEAE Dose Interruption to IP | 221 | 125
  TEAE Leading to Death | 2 | 2
  >=1 Related TEAE Leading to Death | 2 | 2

4. Secondary Outcome: The Number of Participants With Clinical Chemistry Laboratory-Detected Abnormalities (Grade 3-4)
Description: The number of participants with grade 3-4 laboratory abnormalities in selected clinically significant parameters. Grades for chemistry parameters were coded using National Cancer Institute Common Terminology Criteria for Adverse Events (Grade 3= severe, Grade 4= life-threatening).
Time Frame: From day 1 of study drug up to 28 days after the last dose of study drug, or the treatment discontinuation date, whichever was later (up to approximately 37 weeks).
Population: All treated participants with at least one post-baseline value and received at least one dose of investigational product (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel and Gemcitabine | Gemcitabine
Number analyzed (Participants) | 421 | 416
Participants
  Alkaline phosphatase | 7 | 3
  Alanine aminotransferase | 9 | 3
  Aspartate aminotransferase: number analyzed (Participants) | 420 | 416
  Aspartate aminotransferase | 9 | 2
  Bilirubin | 0 | 1

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 94 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 46 weeks)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Nab-Paclitaxel and Gemcitabine | Gemcitabine
All-Cause Mortality (participants affected / at risk) | 285/432 | 297/434
Serious Adverse Events (participants affected / at risk) | 181/429 | 96/423
Other Adverse Events (participants affected / at risk) | 426/429 | 407/423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel and Gemcitabine (N=429) | Gemcitabine (N=423)
Anaemia (Blood and lymphatic system disorders) | 12 | 6
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 3
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 2
Atrial thrombosis (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 4
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 2
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 4
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Anastomotic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Internal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Jejunal perforation (Gastrointestinal disorders) | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 3
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 8 | 0
Asthenia (General disorders) | 4 | 1
Chills (General disorders) | 2 | 2
Fatigue (General disorders) | 7 | 0
General physical health deterioration (General disorders) | 2 | 0
Generalised oedema (General disorders) | 1 | 3
Impaired healing (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 5 | 3
Peripheral swelling (General disorders) | 0 | 1
Polyserositis (General disorders) | 1 | 0
Pyrexia (General disorders) | 29 | 24
Systemic inflammatory response syndrome (General disorders) | 1 | 3
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 4 | 3
Cholangitis acute (Hepatobiliary disorders) | 3 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 2 | 0
Abdominal infection (Infections and infestations) | 4 | 0
Appendicitis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Biliary tract infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 8 | 5
Cholera (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 3 | 0
Colonic abscess (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 2
Device related infection (Infections and infestations) | 4 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 2 | 0
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 1 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 9 | 1
Infectious colitis (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 3 | 0
Lung infection (Infections and infestations) | 2 | 0
Neutropenic sepsis (Infections and infestations) | 2 | 0
Pancreatic abscess (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 9 | 6
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 12 | 5
Septic shock (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 7 | 2
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 2
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Electrocardiogram repolarisation abnormality (Investigations) | 0 | 1
Liver function test increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 4 | 1
Device occlusion (Product Issues) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 1
Embolism (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 2 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 5 | 3
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel and Gemcitabine (N=429) | Gemcitabine (N=423)
Anaemia (Blood and lymphatic system disorders) | 179 | 142
Leukopenia (Blood and lymphatic system disorders) | 84 | 72
Neutropenia (Blood and lymphatic system disorders) | 263 | 230
Thrombocytopenia (Blood and lymphatic system disorders) | 94 | 85
Abdominal pain (Gastrointestinal disorders) | 119 | 87
Abdominal pain upper (Gastrointestinal disorders) | 35 | 40
Constipation (Gastrointestinal disorders) | 114 | 89
Diarrhoea (Gastrointestinal disorders) | 242 | 125
Dyspepsia (Gastrointestinal disorders) | 21 | 24
Flatulence (Gastrointestinal disorders) | 23 | 27
Nausea (Gastrointestinal disorders) | 231 | 192
Stomatitis (Gastrointestinal disorders) | 81 | 24
Vomiting (Gastrointestinal disorders) | 122 | 77
Asthenia (General disorders) | 95 | 49
Chills (General disorders) | 38 | 23
Fatigue (General disorders) | 233 | 203
Influenza like illness (General disorders) | 27 | 25
Oedema peripheral (General disorders) | 162 | 108
Peripheral swelling (General disorders) | 22 | 16
Pyrexia (General disorders) | 171 | 115
Urinary tract infection (Infections and infestations) | 29 | 20
Alanine aminotransferase increased (Investigations) | 42 | 33
Aspartate aminotransferase increased (Investigations) | 31 | 21
Blood alkaline phosphatase increased (Investigations) | 23 | 17
Neutrophil count decreased (Investigations) | 23 | 32
Weight decreased (Investigations) | 52 | 22
Decreased appetite (Metabolism and nutrition disorders) | 143 | 84
Dehydration (Metabolism and nutrition disorders) | 28 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 34 | 28
Hypokalaemia (Metabolism and nutrition disorders) | 55 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 68 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 44
Bone pain (Musculoskeletal and connective tissue disorders) | 23 | 15
Muscular weakness (Musculoskeletal and connective tissue disorders) | 25 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 57 | 29
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 | 33
Dizziness (Nervous system disorders) | 64 | 34
Dysgeusia (Nervous system disorders) | 86 | 36
Headache (Nervous system disorders) | 65 | 66
Neuropathy peripheral (Nervous system disorders) | 112 | 26
Paraesthesia (Nervous system disorders) | 39 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 144 | 16
Polyneuropathy (Nervous system disorders) | 23 | 6
Anxiety (Psychiatric disorders) | 34 | 38
Insomnia (Psychiatric disorders) | 64 | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 61 | 51
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 65 | 50
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 76 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 | 18
Alopecia (Skin and subcutaneous tissue disorders) | 252 | 52
Pruritus (Skin and subcutaneous tissue disorders) | 37 | 20
Rash (Skin and subcutaneous tissue disorders) | 49 | 20
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 35 | 20
Hypertension (Vascular disorders) | 35 | 49
Hypotension (Vascular disorders) | 30 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT01964430/Prot_002.pdf
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT01964430/SAP_001.pdf